CLINICAL TRIAL: NCT00330993
Title: Oral Mifepristone and Buccal Misoprostol Administered Simultaneously for Abortion Through 63 Days Gestation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0601001
Record Dates: First submitted 2006-05-26; First posted 2006-05-29 (Estimated); Last update posted 2007-01-25 (Estimated); Status verified 2006-09

CONDITIONS: Abortion, Induced
Keywords: mifepristone; misoprostol; medical abortion; buccal administration
MeSH Terms: interventions — Mifepristone; Misoprostol

INTERVENTIONS:
Drug: mifepristone, misoprostol

SUMMARY:
HYPOTHESIS: For women with pregnancies at <49, 50-56, and 57-63 days gestation who receive mifepristone 200 mg orally and misoprostol 800 mcg buccally at the same time, the complete abortion rate 24 hours after misoprostol administration will be 90% (95% CI 78%, 97%) within each gestational age group.

This is a prospective clinical trial. Women will be enrolled such that 40 women are in each of three gestational age ranges: ≤49, 50-56, and 57-63 days gestation on the day treatment is initiated. Once a gestational age range includes 40 subjects, enrollment in that group will be closed. Subjects will swallow mifepristone 200 mg and then place four 200 µg misoprostol tablets between the check and gum (2 tablets on each side). The women will be instructed to keep the tablets in place for 30 minutes; any remaining portions of the tablets will be swallowed after this time. Participants will follow-up 24 hours after receiving the misoprostol. Vaginal ultrasonography will be performed to assess for expulsion of the gestational sac. Women who have not aborted by the first follow-up visit will be given a dose of vaginal misoprostol and will return for a follow-up visit in one week. Subjects who have not aborted by the two-week follow-up will be offered a surgical abortion. At each visit, data will be collected on bleeding, cramping, other side effects, and medication use.

DETAILED DESCRIPTION:
1. TELEPHONE SCREEN:

   Initial contact will be by a phone call (or, rarely, a drop-in visit) initiated by a potential study participant. A member of the research staff will advise the potential participant of the study rationale, protocol, risks, benefits, and visit schedule. We request a waiver of the requirement to obtain signed informed consent for the screening process, which will usually take place over the phone. We believe we meet the criteria for the use of this waiver because the screening procedure presents no more than minimal risk of harm to the subjects and involves no procedures for which written consent is normally required outside of the research context. The information obtained during the screening phone call is the same type of information that would be collected on patients setting up an appointment for an abortion. The telephone script and screen are included in Attachment 2. If the subject does not meet inclusion criteria, the information collected during the screening process will be destroyed. Potential subjects interested in participation will be scheduled for a screening visit.

   Each subject will undergo a minimum of 3 visits all of which will be performed in the Family Planning Research Office at Magee-Womens Hospital. She will also receive a minimum of 3 follow-up telephone calls. Those subjects who do not pass the pregnancy by the first follow-up visit will be scheduled for return visits as indicated on the Study Flow Sheet (see attachment) and described below.
2. SCREENING AND ENROLLMENT: Visit length 1 ½ hours.

   1. After obtaining consent for a screening ultrasound evaluation, a transvaginal and a transabdominal ultrasound examination will be performed to ascertain gestational age. The transvaginal ultrasound results will be used to confirm gestational age and document an intrauterine gestation for the study protocol. Vaginal ultrasound to confirm estimated gestational age (EGA) will use the following criteria:

      * EGA (days) = mean sac diameter + 3025
      * EGA (days) = embryonic pole + 4226
      * Mean sac diameter ([length + width + depth]/3) should be used only when no embryonic pole is present.
      * If the ultrasound EGA is different from LMP EGA by 4 days or more, then the ultrasound EGA should be used as the study EGA.
   2. Written informed consent will be obtained at the screening visit prior to any research activities. The investigator or one of the co-investigators, who are physicians, will sign the informed consent document.
   3. After obtaining informed consent, a medical history and initial laboratory tests (hemoglobin and blood type) will be obtained. If the pelvic examination is normal, the endovaginal ultrasound confirms that the gestational age will be less than 63 days on the day of the mifepristone administration, and the laboratory tests satisfy the entry criteria, the subject will be asked to participate in the study.
   4. A HIPAA compliant "Release of Medical Records" form will be signed to allow future access to medical records related to any care provided during the study by another health care provider.
3. VISIT 1: The subject will return prior to reaching 64 days gestation. This day will be considered Study Day 1. Visit length 30 minutes.

   1. The research staff will administer a pre-study questionnaire. The subject will complete a Visual Analogue Scale (VAS) assessment.
   2. Eligibility criteria will be reviewed and, if indicated by a history of bleeding since screening, a vaginal ultrasound will be performed.
   3. A licensed clinician will distribute the medications after completion of the questionnaire. The medications will be kept in a locked file in the research office and a log will be generated to track medication usage, lot numbers, and expiration dates. All subjects will take the mifepristone and misoprostol in front of the research clinician.

      * She will receive mifepristone 200 mg orally and swallow the tablet in front of one of the researchers. THE SUBJECT CANNOT RECEIVE THE MIFEPRISTONE UNTIL A MINIMUM OF 24 HOURS AFTER COMPLETION OF THE INFORMED CONSENT.
      * Within 5 minutes of mifepristone administration, the subject will be given four 200 µg tablets of misoprostol to place between the cheek and gum (2 on each side) and to allow them to remain in that location for 30 minutes. After this time lapse, any remaining tablets will be swallowed. The subject will not need to wait in the office during the 30 minutes.
   4. The subject will receive a prescription for codeine (30 mg) or hydrocodone (5 mg), #20 and an instruction sheet with the phone numbers to call if she has any questions or problems.
   5. Rh-immune globulin will be administered if she is Rh-negative.
   6. The subject will be scheduled for follow-up 24 ± 1 hours after administration of the misoprostol.
4. VISIT 2: 24 ± 1 hours after misoprostol administration. Visit length 1 hour.

   1. Endovaginal and abdominal ultrasound examinations will be performed.

      * If the vaginal ultrasound examination demonstrates a gestational sac, the subject will receive a "rescue" dose of vaginal misoprostol (four 200 µg tablets of misoprostol), which will be placed by the clinician. A follow-up appointment will be scheduled for study Day 15 (range Day 13-17)
      * If the vaginal ultrasound does not demonstrate a sac the abortion will be considered complete and telephone follow-up contacts will be the only scheduled evaluations from this point forward.
   2. All subjects will complete a post-study VAS, which will take about 5 minutes to complete.
5. TELEPHONE FOLLOW-UP #1: Study Day 8 (range Day 6-10). Call length 10 minutes. Subjects will be contacted to assess their clinical status including bleeding, cramping, and medication requirements. If necessary, based on the subject's responses, appointments for evaluation by a clinician will be made at that time.
6. VISIT 3/TELEPHONE FOLLOW-UP #2: Study Day 15 (range Day 13-17). Visit length (if required) 1 hour, call length 10 minutes)

   1. Subjects who had expelled the gestational sac as based on prior ultrasound examination will receive telephone follow-up to assess their clinical status. Appointments for evaluation by a clinician will be made as necessary. A post-study acceptability questionnaire will be performed with these subjects over the telephone, which will take about 5 minutes to complete.
   2. Subjects who had not expelled the gestational sac on prior examination will return to the office for this visit. Endovaginal and abdominal ultrasounds will be performed.

      * If the vaginal ultrasound shows an intrauterine gestation with embryonic cardiac activity, the subject will be offered and advised to have a surgical abortion to be done as soon as possible. After the D&C, the subject will complete a 5-minute post-study acceptability questionnaire. She will also have a telephone follow-up on Study Day 36.
      * If the vaginal ultrasound shows the gestational sac to be present without embryonic cardiac activity, the subject may have a D&C and complete the acceptability questionnaire or can pursue expectant management and return on Study Day 36 (range Day 32-40).
      * If the vaginal ultrasound demonstrates absence of the gestational sac, she will complete a post-study acceptability questionnaire at the end of her visit which will take about 5 minutes to complete and all further follow up will be performed by telephone.
7. VISIT 4/TELEPHONE FOLLOW_UP #3: Study Day 36 (range Day 32-40). Visit length (if required) 30 minutes-1 hour, call length 10 minutes.

   1. Subjects who had expelled the gestational sac as based on prior ultrasound examination or who had a D&C will receive telephone follow-up to assess their clinical status. Appointments to be evaluated by a clinical will be made as necessary.
   2. If the subject must return for this visit, endovaginal and abdominal ultrasound examinations will be performed. If the vaginal ultrasound shows the gestational sac to still be present, the patient will be offered a surgical abortion.
   3. At the completion of the surgical abortion or if the ultrasound demonstrates absence of a sac, a 5-minute post-study acceptability questionnaire will be performed.
8. OTHER

   1. The subject will be questioned at each visit regarding side effects experienced from the medications, bleeding and cramping, pain medication required, and other medications used since the last visit.
   2. If the subject does not return for a scheduled visit, she should be telephoned to reschedule the visit. If the patient is unable to return for her follow-up, the required information regarding bleeding history, medications, medication side effects, and questionnaire answers can be obtained over the phone. If the subject is unable to be reached by phone within two weeks of her scheduled visit, a certified letter must be sent indicating her need to return. Subjects will be considered lost to follow-up only if the final visit is not completed by the time the study is closed.
   3. If the subject fails to return for her Visit 2, but returns at some later time during her study participation period and is found to have a retained gestational sac or continuing pregnancy on ultrasound, she may receive an additional vaginal dose of misoprostol (4 tablets; up to Study Day 12) or be offered a D&C (at any time).
   4. The subject will be counseled not have intercourse or drink alcohol until the completion of the abortion is confirmed.
   5. Contraceptive counseling will be performed throughout the study. A method of contraception should be instituted after the abortion has occurred and before the subject resumes sexual activity.
   6. Endovaginal ultrasound may be performed at any time other than what is required by the protocol if felt to be necessary by the clinician.
   7. Standard suction curettage will be performed for continuing pregnancy at visit 3 or persistent sac at visit 4, uterine hemorrhage, or incomplete abortion.

ELIGIBILITY:
Inclusion Criteria:Healthy females: 1) 18 years of age or older, 2) requesting an elective termination of pregnancy by medical abortion, 3) with an intrauterine pregnancy no more than 63 days gestation on the day of mifepristone administration as documented by endovaginal ultrasound, 4) willing and able to sign informed consent, 5) willing to comply with the study protocol and visit schedule, 6) willing to have a surgical abortion/D&C if indicated, and 7) with easy and ready access to a telephone.

-

Exclusion Criteria:1) ultrasound evidence at the evaluation(s) prior to mifepristone treatment of an early pregnancy failure, 2) contraindication to mifepristone (known allergy to mifepristone, chronic corticosteroid administration, adrenal disease), 3) contraindication to misoprostol (glaucoma, mitral stenosis, sickle cell anemia, poorly controlled seizure disorder, or known allergy to prostaglandin), 4) known or suspected extrauterine pregnancy, 5) known or suspected pelvic infection, 6) hemoglobin <10 mg/dL, 7) known clotting defect or receiving anticoagulants, 8) cardiovascular disease (angina, valvular disease, arrhythmia, or cardiac failure), 9) current breastfeeding, 10) pregnancy with an IUD in situ, 11) current use of any experimental drug, 12) suspected or confirmed endometrial arteriovenous malformation, 13) active oral herpes lesions per subject report, 14) prior participation in this research study, or 15) current participation in another research study that, in the opinion of the investigator, would interfere with the conduct of this study.

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-03; Study Completion 2006-08

PRIMARY OUTCOMES:
To determine the complete abortion rate, at 24 hours after misoprostol administration, when using mifepristone 200 mg orally and misoprostol 800 mcg buccally simultaneously in women at <49, 50-56, and 57-63 days gestation.

SECONDARY OUTCOMES:
To compare the complete abortion rates, at 24 hours after misoprostol administration, by gestational age (up to and including 49, from 50-56, and 57-63 days gestation) with this medical abortion regimen.
To determine the complete medical abortion rate at approximately 14 days after treatment, among those women who receive a second dose of misoprostol.
To assess side effects (i.e. nausea, vomiting) and pain medication use after treatment.
To assess the acceptability of this medical abortion regimen.
To compare the accuracy of transvaginal and abdominal ultrasonography in gestational age dating and treatment failure in this cohort.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia A. Lohr, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Office of Family Planning Research, Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States